CLINICAL TRIAL: NCT03085537
Title: Effectiveness Monitoring of Home Non-invasive Mechanical Ventilation by Pressure and Flow-time Signals Analysis Integrated on Digital Diagnosis Platform.
Brief Title: Effectiveness Monitoring of Home Non-invasive Mechanical Ventilation by Digital Diagnosis Platform
Acronym: PRE-HVNI
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Manel Lujan-Torne, Lung specialist doctor, Corporacion Parc Tauli
Other Study IDs: 13/088
Record Dates: First submitted 2017-03-03; First posted 2017-03-21 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2017-03

CONDITIONS: Neuromuscular Diseases; Obesity Hypoventilation Syndrome; Lung Disease, Restrictive
Keywords: home monitoring; Non-invasive mechanical ventilation
MeSH Terms: conditions — Neuromuscular Diseases; Obesity Hypoventilation Syndrome; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
The main objective will be to determine the effectiveness of home non-invasive ventilation by flow-time and time-pressure curves analysis in a cohort of patients with this treatment by digital diagnosis platform.

DETAILED DESCRIPTION:
A multicenter study with observational prospective design will be implemented on 3 spanish hospitals in Barcelona. Inclusion criteria will be equivalent sample size of patients with restrictive lung disease, neuromuscular pathology and hypoventilation-obesity.

Digital diagnosis platform will be used to incorporate and unify signals of different medical devices: a pneumotachograph on branch ventilator that captures pressure and flow-time signals, inductance plethysmography used to like a patient effort sensor and portable pulse oximeter recordings. Nocturnal polygraphic or polysomnographic tracings performed and recorded on sites will be processed systematically by main asynchronies diagnosis algorithms between patient and ventilator. These algorithms providing global and fractionated asynchronies count based on time, leaks or saturation criteria which will be used to compared effective ventilation phases and phases with nocturnal desaturations. Therefore, prevalence and asynchronies model on home NIV can be determine establishing the correlation between desaturation phases and respiratory events and identifying minimum tolerable leak level to keep adequate ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Home non-invasive mechanical ventilation and clinical stability at least of 6 months ( no acute episode with admission on 2 months before)
* Mean Ventilator compliance > 4 h/ per night on screening visit
* Signed informed consent form previously

Exclusion Criteria:

* Ventilation with oxygen join system.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by restrictive lung disease, neuromuscular disorders or hypoventilation-obesity with home non-invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Asynchronies Index | One week after screening visit if the subject comply inclusion criteria. Asynchronies analysis will be performed once (cross-sectional design) by nocturnal polygraphy on site during one night
  Number of respiratory events registered automatically by digital diagnosis platform

SECONDARY OUTCOMES:
Leaks | One week after screening visit if the subject comply inclusion criteria. leaks analysis will be performed once (cross-sectional design) by nocturnal polygraphy on site during one night
  Presence or not of intencionals and unintencionals leaks recorded
Oxygen saturation | One week after screening visit if the subject comply inclusion criteria. Oxygen saturation analysis will be performed once by nocturnal polygraphy once (cross-sectional design) on site during one night
  Measure by pulsy oxymetry (%)
Demographics parameters- age | screening visit
  age in years
Demographics parameters- sex | screening visit
  sex: man or woman
Pathology indication | screening visit
  asociated with starting mechanical ventilation
PaCO2 | screening visit
  PaCo2 measured by blood gas test (mmHg) < 45
Pittsburgh Sleep Quality Index. (PSQI) | screening visit
  questionaire of sleep quality with ventilation.
Mode Ventilator | recorded date on screening visit
  pressure or volume controlled modes. select the option at ventilator setings
Interfaces | recorded date on screening visit
  kind of mask using between the patient and ventilator. Total face mask, nasal mask, oro-nasal mask depend of patient characteristics
Tube | recorded date on screening visit
  Kind of tuve, simple or doublé between patient and ventilator
Antyrebreathing system | recorded date on screening visit
  Kind of system that avoid rebreathing CO2: acitve valve, leak controlled mask, leak controlled tube or double circuit
Compliance ventilator | recorded date on screening visit
  complying or not mínimum hours to recruiting (4h)

CONTACTS AND LOCATIONS:
Overall Officials: Manel Lujan, Principal Investigator — Corporation PT
Locations (3):
- Spain (3):
  - Hospital universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporación Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Vall d´Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided